CLINICAL TRIAL: NCT07318506
Title: Effects of Staged Adapted Inclusions in Infant Cereals on Oral-motors Patterns of 6-24 Month-old Children
Acronym: ICONIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2506INF
Record Dates: First submitted 2025-11-26; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Infant and Young Child Feeding
MeSH Terms: interventions — Fumigant 93

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- A, B, E, C, D (Other): Cross-over sequence. Test product E is not applicable for 6-8 months and 18-24 months age group.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- B, C, A, D, E (Other): Cross-over sequence starting by test product B. Test product E is not applicable for 6-8 months and 18-24 months age group.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- C, D, B, E, A (Other): Cross-over sequence.Test product E is not applicable for 6-8 months and 18-24 months age group.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- D, E, C, A, B (Other): Cross-over sequence. Test product E is not applicable for 6-8 months and 18-24 months age group.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- E, A, D, B, C (Other): Cross-over sequence. Test product E is not applicable for 6-8 months and 18-24 months age group.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- D, C, E, B, A (Other): Cross-over sequence. Test product E is not applicable for 6-8 months and 18-24 months age group.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- E, D, A, C, B (Other): Cross-over sequence. Test product E is not applicable for 6-8 months and 18-24 months age group.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- A, E, B, D, C (Other): Cross-over sequence. Test product E is not applicable for 6-8 months and 18-24 months age group.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- B, A, C, E, D (Other): Cross-over sequence. Test product E is not applicable for 6-8 months and 18-24 months age group.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E
- C, B, D, A, E (Other): Cross-over sequence. Test product E is not applicable for 6-8 months and 18-24 months age group.
  Interventions: Other: A; Other: B; Other: C; Other: D; Other: E

INTERVENTIONS:
Other: A — Control: base infant rice-based cereal with no added sugar
Other: B — Test product: base infant rice-based cereal with age appropriate inclusions. Inclusion type 1 for 6-8 months age group; type 4 for 8-12 months age group; type 4 for 12-18 months age group; type 9 for 18-24 months age group.
Other: C — Test product: base infant rice-based cereal with age appropriate inclusions. Inclusion type 2 for 6-8 months age group; type 5 for 8-12 months age group; type 6 for 12-18 months age group; type 10 for 18-24 months age group.
Other: D — Test product: base infant rice-based cereal with age appropriate inclusions. Inclusion type 3 for 6-8 months age group; type 6 for 8-12 months age group; type 8 for 12-18 months age group; type 11 for 18-24 months age group.
Other: E — Test product: base infant rice-based cereal with age appropriate inclusions. Inclusion type 7 for 8-12 months and 18-24 months age groups. Not applicable for 6-8 months and 18-24 months age group.

SUMMARY:
The purpose of this study is to define the effects of different inclusions in infant cereals on the adaptation of oral motor behavior and skills displayed at a given age.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 6 months (182 days) to 24 months (730 days) of age (from enrollment to last visit):

   1.1. [182-242]-days of age from V1 to last visit for the 6-8-month-old age group 1.2. [243-364]-days of age from V1 to last visit for the 8-12-month-old age group 1.3. [365-547]-days of age from V1 to last visit for the 12-18-month-old age group 1.4. [548-730]-days of age from V1 to last visit for the 18-24-month-old age group
2. Singleton, full-term infants (≥ 37 completed weeks of gestation), with a birth weight of ≥ 2.5 kg and ≤ 4.5 kg.
3. Healthy children based on medical history as reported by parent(s) / LAR(s).
4. Sit upright with or without support (such as, sitting with back against a chair or while being held) as reported by parent(s) / LAR(s)
5. Keep head steady when in a supported position
6. Have already started complementary feeding as recommended by their health care professional (have started solid food beyond breastmilk or infant formula)
7. Written informed consent is obtained from at least one parent(s) / LAR(s).
8. Parent(s) / LAR(s) must be able to provide evidence of parental authority and identity.
9. Parent(s) / LAR(s) must understand the informed consent and other study documents.
10. Parent(s) / LAR(s) are willing and able to fulfill the requirements of the study protocol within the study timeframe.

Exclusion Criteria:

* 1. Infant's parents or LARs have not reached legal age of majority (18 years) 2. Children with history of oral/facial malformations or surgery (i.e. cleft lip, cleft palate, tongue-tie/ankyloglossia), or history of tube feeding for any reason.

  3. Children with any chronic illness, congenital malformations (e.g., esophageal or intestinal atresia), surgical sequela (e.g., short bowel syndrome), gastroesophageal reflux disease, behavioral disorders, neurodevelopmental delay or illness that impacts feeding. [children with an acute illness, such as a cold, gastroenteritis etc. can be included but can only attend the visits once they have recovered].

  4. Children with feeding or swallowing difficulties/disorders, history of choking, or at high risk of choking.

  5. Child or sibling(s) who has known or suspected food allergy or intolerance, such as cows' milk protein allergy, celiac disease, lactose intolerance, soy allergy, fish allergy, or any other suspected or confirmed food allergies or intolerance.

  6. Children with undernutrition as determined by age-group weight threshold (based on parental reports): weight at [6-8[month < 6 kg; weight at [8-12[months: < 6.5 kg; weight at [12-18[months: < 7.5 kg; weight at [18-24] months: < 8.5 kg.

  7. Child is currently participating in or has participated in another intervention clinical study that impacts study outcomes within 4 weeks prior to enrolment or has participated in another age group of this study.

  8. Family or hierarchical relationships with the research team members.

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 153 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Effects of different inclusions in infant cereals on the number of chews according to the age group. | Immediately after the product intake
  Define the change in number of chews observed during consumption of infant cereals with or without different inclusions based on manual video coding

SECONDARY OUTCOMES:
Impact of different inclusions on oral motor movement during consumption of infant cereals according to age group. | Immediately after the product intake
  Comparer chewing duration extracted from video manual coding and the Baby FaceReader automatically calculated metrics between products with different textures for each age group.
Impact of different inclusions on oral motor movement during consumption of infant cereals according to age group. | Immediately after the product intake
  Comparer chewing rate extracted from video manual coding and the Baby FaceReader automatically calculated metrics between products with different textures for each age group.
Impact of different inclusions on oral motor movement during consumption of infant cereals according to age group. | Immediately after the product intake
  Comparer the observation of tongue lateral movements extracted from video manual coding and the BabyFaceReader automatically calculated metrics between products with different textures for each age group, using a 3 points categorical scale.
Impact of different inclusions on oral motor movement during consumption of infant cereals according to age group. | Immediately after the product intake
  Comparer the observation of rotary chewing motions extracted from video manual coding and the Baby FaceReader automatically calculated metrics between products with different textures for each age group, using a 3 points categorical scale.
Associations between inclusion properties and oral motor movement according to age group. | Immediately after the product intake
  Identify specific correlation between product texture sensorial caracteristics data and number of chews for each age group, using Partial Least Squares Regression.
Associations between inclusion properties and oral motor movement according to age group. | Immediately after the product intake
  Identify specific correlation between product texture mechanical caracteristics data and number of chews for each age group, using Partial Least Squares Regression.
Impact of inclusions on food acceptance during consumption of infant cereals according to age group. | Immediately after the product intake
  Comparer between product textures and according to the age group time to consume 5 spoons
Impact of inclusions on food acceptance during consumption of infant cereals according to age group. | Immediately after the product intake
  Comparer between product textures and according to the age group time to consume each individual spoon
Impact of inclusions on food acceptance during consumption of infant cereals according to age group. | Immediately after the product intake
  Comparer between product textures and according to the age group occurrence of positive and negative behaviors per session
Impact of inclusions on food liking during consumption of infant cereals according to age group. | Immediately after the product intake
  Comparer parents reported liking between product textures for each age group based on the score of liker scale responses (dislike extremely score to like extremely score).

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Instituto DYM S.A., Barcelona
  - Institute of Agrochemistry & Food Technology CSIC, Valencia

IPD SHARING:
Plan to Share IPD: No